CLINICAL TRIAL: NCT02143609
Title: Patients With Chronic Obstructive Pulmonary Disease at Altitude - Effect of Nocturnal Oxygen Therapy on Exercise Performance
Brief Title: Patients With Chronic Obstructive Pulmonary Disease at Altitude - Effect of Nocturnal Oxygen on Exercise Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0088V2A3
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; lung
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Active Comparator): oxygen administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Interventions: Drug: oxygen; Drug: sham oxygen (room air)
- Sham oxygen (Placebo Comparator): sham oxygen (room air) administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Interventions: Drug: oxygen; Drug: sham oxygen (room air)

INTERVENTIONS:
Drug: oxygen — Nocturnal nasal oxygen during stay at 2048 m
  Other Names: Nocturnal oxygen via nasal cannula, 3 L/min, at 2048 m
Drug: sham oxygen (room air) — Sham oxygen (room air) via nasal cannula, 3 L/min, at 2048 m
  Other Names: Nocturnal nasal room air during stay at 2048 m

SUMMARY:
The purpose of this study is to investigate the effect of nocturnal oxygen therapy during a stay at moderate altitude on exercise performance of patients with chronic obstructive lung disease.

DETAILED DESCRIPTION:
Patients with moderate to severe COPD living below 800 m, will be recruited to participate in a randomized cross-over field trial evaluating the hypothesis that exercise capacity during a 2 day sojourn at moderate altitude is improved by nocturnal oxygen therapy via a nasal cannula. Outcomes will be assessed during 2 days in Zurich (490 m, low altitude baseline), and during 2 days at St. Moritz Salastrains (2048 m).

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease (COPD), GOLD grade 2-3
* residents at low altitude (<800 m)

Exclusion Criteria:

* unstable condition, COPD exacerbation
* mild (GOLD 1) or very severe COPD (GOLD 4)
* requirement for oxygen therapy at low altitude residence
* hypoventilation
* pulmonary hypertension
* more than mild or unstable cardiovascular disease
* use of drugs that affect respiratory center drive
* internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day), inability to perform 6 min walk test.
* previous intolerance to moderate altitude (<2600m).
* exposure to altitudes >1500m for >2 days within the last 4 weeks before the study.
* pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
6 min walk distance | Day 2 at 2048 m
  Difference in the distance walked in 6 min between the oxygen and sham oxygen period

SECONDARY OUTCOMES:
6 min walk distance | day 3 at 2048 m
  Difference in the distance walked in 6 min between the oxygen and sham oxygen period
Arterial blood gas analysis | Day 2 at 2048 m
  Difference in arterial oxygen partial pressure, carbon dioxide partial pressure, and pH
Spirometry | Day 2 at 2048 m
  Difference in spirometric variables between the oxygen and sham oxygen period
Perceived exertion | Day 2 at 2048 m
  Difference in perceived exertion rated with the BORG CR10 scale at the end of the 6 min walk
Perceived exertion | Day 3 at 2048 m
  Difference in perceived exertion rated with the BORG CR10 scale at the end of the 6 min walk
Severe hypoxemia | Day 1 to 3 at 2048 m
  Number of participants in whom arterial oxygen saturation measured by pulse oximetry is less than 75% for more than 30 min during the oxygen and sham oxygen treatment periods at 2028 m.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland